CLINICAL TRIAL: NCT04911166
Title: Phase I Trial of Atezolizumab and Interleukin-12 Gene Therapy in Metastatic Non-Small Cell Lung Cancer With Progression on First-Line Immunotherapy With or Without Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, Associate Professor of Clinical Medicine in Oncology, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00026826
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Atezolizumab; Gene therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: This is a Phase I study evaluating the safety of atezolizumab in combination with ADV/IL-12 gene therapy in patients with metastatic NSCLC whose disease has progressed on first-line immunotherapy with or without chemotherapy. Approximately 16 patients will be enrolled on the study. ADV/IL-12 will be intratumorally injected on Day 0 of the study. The starting dose of ADV/IL-12 will be 5 × 1011 vp. Starting on Day 2 of the study, atezolizumab will be administered at 1200 mg IV Q3W for 2 cycles. Patients with SD or better after completion of 2 cycles of atezolizumab will continue to receive atezolizumab Q3W until disease progression, unacceptable toxicity, or up to 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and Interleukin-12 Gene Therapy (Experimental)
  Interventions: Combination Product: Atezolizumab and Interleukin-12 Gene Therapy

INTERVENTIONS:
Combination Product: Atezolizumab and Interleukin-12 Gene Therapy — To determine the safety and tolerability of the atezolizumab and ADV/IL-12 gene therapy combination in patients with metastatic NSCLC who have disease progression after a prior line of either single agent immunotherapy or a regimen of chemoimmunotherapy.

SUMMARY:
This is a Phase I study evaluating the safety of atezolizumab in combination with ADV/IL-12 gene therapy in patients with metastatic non-small cell lung cancer (NSCLC) whose disease has progressed on first-line immunotherapy with or without chemotherapy.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety of atezolizumab in combination with adenoviral-mediated interleukin-12 (ADV/IL-12) gene therapy in patients with metastatic non-small cell lung cancer (NSCLC) whose disease has progressed on first-line immunotherapy with or without chemotherapy. Approximately 16 patients will be enrolled on the study. The primary endpoint will be the safety of the atezolizumab and ADV/IL-12 gene therapy combination and will be determined using the Bayesian model averaging-continual reassessment method (BMA-CRM). ADV/IL-12 will be intratumorally injected on Day 0 of the study. The starting dose of ADV/IL-12 will be 5 × 1011 vp. ADV/IL-12 dose level will de-escalate based on Dose Limiting Toxicity (DLT) occurrence: dose level -1, 3 × 1011 vp and dose level -2, 1 × 1011 vp. The starting dose, based on the dose range explored in prior studies, is expected to have activity and dosing changes are only in place in the event that toxicity is demonstrated. Starting on Day 2 of the study, atezolizumab will be administered at 1200 mg IV every 3 weeks (Q3W) for 2 cycles. Patients with stable disease or better after completion of 2 cycles of atezolizumab will continue to receive atezolizumab Q3W until disease progression, unacceptable toxicity, or up to 12 months.

ELIGIBILITY:
INCLUSION CRITERIA

Patients must meet the following criteria for study entry:

1. Signed informed consent form.
2. Male or female.
3. Age ≥ 18 years at time of signing informed consent form.
4. Ability to comply with the study protocol, in the investigator's judgment.
5. Histologically or cytologically confirmed metastatic NSCLC.
6. Disease progression on first-line immunotherapy with or without chemotherapy (chemoimmunotherapy [e.g., carboplatin/pemetrexed/pembrolizumab] or single-agent pembrolizumab in PD-L1-expressing tumors). Patients with National Comprehensive Cancer Network recommended targeted mutations who have failed FDA-approved targeted therapies for these aberrations will be eligible for enrollment in the study.
7. Measurable disease per RECIST v1.1. Previously irradiated lesions can be considered as measurable disease only if progressive disease (PD) has been unequivocally documented at that site since radiation.
8. Accessible tumor for ADV/IL-12 administration (a lesion safely accessible by an image guided biopsy or bronchoscopy) .
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 3).
10. Life expectancy ≥6 months.
11. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 28 days prior to initiation of study treatment:

    * Absolute neutrophil count (ANC) ≥1500/µL without granulocyte colony-stimulating factor support within 14 days of assessment)
    * Lymphocyte count ≥ 500/µL
    * WBC count >2,500/µL and <15,000/µL
    * Platelet count ≥100,000/µL (without transfusion within 7 days of assessment)
    * Hemoglobin ≥9 g/dL (without transfusion within 7 days of assessment)
    * AST, ALT, and alkaline phosphatase (ALP) ≤2.5 × upper limit of normal (ULN), with the following exceptions: Patients with documented liver metastases: AST and ALT ≤5 × ULN Patients with documented liver or bone metastases: ALP ≤5 × ULN
    * Serum bilirubin ≤1.5 × ULN with the following exception:

    Patients with known Gilbert disease: serum bilirubin level ≤3 × ULN
    * Serum creatinine ≤1.8 × ULN
    * For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤1.5 × ULN.
12. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen (i.e. on a stable dose of anticoagulants for a minimum of 2 weeks).
13. Negative human immunodeficiency virus (HIV) test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥200/µL, and have an undetectable viral load.
14. Negative hepatitis B surface antigen (HBsAg) test at screening.
15. Cardiac ejection fraction of ≥45%.
16. ≥4 weeks since any major surgery, completion of radiation therapy, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy).
17. Willing to provide biopsy tissue as required by the study.
18. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below: Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 5 months after the final dose of study treatment. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
19. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below: With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 5 months after the final dose of study treatment. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure.

EXCLUSION CRITERIA

Patients who meet any of the following criteria will be excluded from study entry:

1. History of leptomeningeal disease.
2. Uncontrolled tumor-related pain Patients requiring pain medication must be on a stable regimen at study entry Palliative radiotherapy is allowed to a single painful metastatic site during the study if the patient is otherwise benefitting from the study treatment per the treating physician's judgment.
3. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX®) are allowed.
4. Uncontrolled or symptomatic hypercalcemia (ionized calcium >1.5 mmol/L, calcium >12 mg/dL or corrected serum calcium >ULN).
5. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions: Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   * Rash must cover <10% of body surface area
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
6. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), druginduced pneumonitis, or idiopathic pneumonitis History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
7. Active tuberculosis
8. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease [Appendix 4], myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
9. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
10. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease [COPD] exacerbation) are eligible for the study.
11. Prior allogeneic stem cell or solid organ transplantation.
12. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
13. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab treatment.
14. Current treatment with anti-viral therapy for hepatitis virus B (HBV).
15. Prior treatment with gene vector therapy.
16. Prior active malignancy within the previous 2 years. NOTE: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that have undergone potentially curative therapy are not excluded.
17. Known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
18. Treatment with investigational therapy within 28 days prior to initiation of study treatment.
19. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
20. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha [TNF-α] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions: Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for COPD or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study. Patients may receive systemic glucocorticoids during study treatment to modulate symptoms from an AE of suspected immunologic etiology.
21. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
22. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.
23. Known allergy or hypersensitivity to any component of the ADV/IL-12 formulation.
24. Pregnancy, breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of study treatment Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival plus stable disease after 6 cycles | 12 weeks
  The primary efficacy endpoint will be the progression-free survival (complete response, partial response) plus stable disease after 6 cycles of atezolizumab) of patients treated with atezolizumab and IL-12 gene therapy in metastatic non-small cell lung cancer with progression on first-line immunotherapy with or without chemotherapy.

SECONDARY OUTCOMES:
Overall Survival | 12 weeks
  Overall Survival of patients treated with atezolizumab and IL-12 gene therapy in metastatic non-small cell lung cancer with progression on first-line immunotherapy with or without chemotherapy.
Radiographic response rate | 12 Weeks
  Radiographic response rate of patients treated with atezolizumab and IL-12 gene therapy in metastatic non-small cell lung cancer with progression on first-line immunotherapy with or without chemotherapy
Health-Related Quality-of-Life (HRQOL) | 12 weeks
  Health-related quality-of-life of patients treated with atezolizumab and IL-12 gene therapy in metastatic non-small cell lung cancer with progression on first-line immunotherapy with or without chemotherapy
Patient-reported outcomes (PRO) | 12 weeks
  Patient-reported outcomes (PRO) of patients treated with atezolizumab and IL-12 gene therapy in metastatic non-small cell lung cancer with progression on first-line immunotherapy with or without chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No